CLINICAL TRIAL: NCT00132080
Title: Trial of Pulse Steroid Therapy in Kawasaki Disease (A Trial Conducted by the Pediatric Heart Network)
Brief Title: Trial of Pulse Steroid Therapy in Kawasaki Disease--Pediatric Heart Network
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pediatric Heart Network (Other)
Responsible Party: Lynn Sleeper, ScD, PI, New England Research Institutes
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 241; U01HL068270 (NIH)
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2012-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Infection; Coronary Aneurysm
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Infections; Coronary Aneurysm | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Placebo Comparator): Patients with acute Kawasaki disease
  Interventions: Drug: Steroids

INTERVENTIONS:
Drug: Steroids — This study evaluates the efficacy and safety of pulse steroid therapy, when added to conventional treatment with IVIG plus aspirin, in treatment of children with acute Kawasaki disease.
  Other Names: pulse steroid therapy.

SUMMARY:
The primary endpoint is coronary artery diameter, normalized for body surface area, 5 weeks after randomization. Secondary endpoints include duration of fever, CRP levels, and adverse events.

DETAILED DESCRIPTION:
BACKGROUND:

Kawasaki Disease (KD) is an inflammatory vasculitis of unknown etiology that affects infants and children and can cause coronary artery aneurysms. Standard therapy consists of 2 gm/kg of intravenous immune globulin plus high-dose aspirin in the acute phase, and low-dose aspirin in the convalescent phase. Some children do not respond to this therapy, and some children go on to develop coronary artery aneurysms in spite of aggressive treatment. This led to the design of this randomized controlled trial to compare a single dose of intravenous steroids vs. placebo on the background of standard therapy. Recruitment began in December, 2002 and ended in December, 2004 with nearly 200 patients randomized.

DESIGN NARRATIVE:

This is a randomized controlled trial to compare a single dose of intravenous steroids vs. placebo on the background of standard therapy

ELIGIBILITY:
* Fever persisting at least 4 days and the presence of at least 4 of the following 5 principal features:

  1. Changes in extremities: Acute changes include erythema and edema of hands and feet; Convalescent changes include membranous desquamation of fingertips
  2. Polymorphous exanthema
  3. Bilateral, painless bulbar conjunctival injection without exudates
  4. Changes in lips and oral cavity: Erythema and cracking of lips, strawberry tongue, diffuse injection of oral and pharyngeal mucosae
  5. Cervical lymphadenopathy ( 1.5 cm in diameter), usually unilateral;

OR

* Patients with at least four days of fever and coronary artery disease, defined as either:

  1. Having a z-score in either the proximal right coronary artery or the proximal left anterior descending coronary artery of > 2.5 detected by 2-dimensional echocardiography, as well as:
* For patients under six months of age, at least two principal criteria
* For patients at least six months of age, at least three principal criteria. 2. Meeting Japanese Ministry of Health criteria for coronary aneurysm defined as an internal lumen diameter of >3 mm in children less than 5 years of age or >4 mm in children 5 years of age and older, in either the proximal right coronary artery or the proximal left anterior descending coronary artery and at least one principal criterion.

AND Enrollment within ten days of the onset of illness, with Day 1 defined as the first day of fever AND Informed consent of parents and assent of children who are older than age 7 years and capable of understanding or according to institutional guidelines.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 199 (Actual)
Dates: Start 2002-12; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Compare the effect of IVMP plus IVIG to IVIG alone on coronary artery outcomes | Measured 5 weeks post-randomization

SECONDARY OUTCOMES:
Occurrence of CA aneurysms; individual z scores of the LMCA, proximal RCA, and proximal LAD CA at 1 and 5 weeks; changes in absolute coronary dimensions for all CA segments from baseline to 1 and 5 weeks after randomization | Measured 5 weeks post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Sleeper, ScD., Principal Investigator — New England Research Institutes, Watertown, MA

REFERENCES:
- [Derived] Printz BF, Sleeper LA, Newburger JW, Minich LL, Bradley T, Cohen MS, Frank D, Li JS, Margossian R, Shirali G, Takahashi M, Colan SD; Pediatric Heart Network Investigators. Noncoronary cardiac abnormalities are associated with coronary artery dilation and with laboratory inflammatory markers in acute Kawasaki disease. J Am Coll Cardiol. 2011 Jan 4;57(1):86-92. doi: 10.1016/j.jacc.2010.08.619. PMID 21185506
- [Derived] Sleeper LA, Minich LL, McCrindle BM, Li JS, Mason W, Colan SD, Atz AM, Printz BF, Baker A, Vetter VL, Newburger JW; Pediatric Heart Network Investigators. Evaluation of Kawasaki disease risk-scoring systems for intravenous immunoglobulin resistance. J Pediatr. 2011 May;158(5):831-835.e3. doi: 10.1016/j.jpeds.2010.10.031. Epub 2010 Dec 18. PMID 21168857
- [Derived] Baker AL, Lu M, Minich LL, Atz AM, Klein GL, Korsin R, Lambert L, Li JS, Mason W, Radojewski E, Vetter VL, Newburger JW; Pediatric Heart Network Investigators. Associated symptoms in the ten days before diagnosis of Kawasaki disease. J Pediatr. 2009 Apr;154(4):592-595.e2. doi: 10.1016/j.jpeds.2008.10.006. Epub 2008 Nov 28. PMID 19038400
- [Derived] Newburger JW, Sleeper LA, McCrindle BW, Minich LL, Gersony W, Vetter VL, Atz AM, Li JS, Takahashi M, Baker AL, Colan SD, Mitchell PD, Klein GL, Sundel RP; Pediatric Heart Network Investigators. Randomized trial of pulsed corticosteroid therapy for primary treatment of Kawasaki disease. N Engl J Med. 2007 Feb 15;356(7):663-75. doi: 10.1056/NEJMoa061235. PMID 17301297